CLINICAL TRIAL: NCT06062121
Title: Pilot Study of Motor-cable-driven System for Stroke Wrist and Forearm Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.166
Record Dates: First submitted 2023-08-31; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- motor-cable-driven system (Experimental): Receive motor-cable-driven system
  Interventions: Device: Motor-cable-driven Rehabilitation Robotic System

INTERVENTIONS:
Device: Motor-cable-driven Rehabilitation Robotic System — Subjects will wear the motor-cable-driven system and receive 30 minutes (including preparation time) wrist and forearm robot-assisting exercise

SUMMARY:
The research purpose is to investigate the feasibility of using a motor-cable-driven system for wrist and forearm recovery of hemiplegic subjects suffered from stroke, where assistive force would be generated from cables connected to pulleys and electrical motors. The system may use EMG signal to control the movements.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute and chronic stroke patients (ischemic or hemorrhagic).
* Sufficient cognition to follow simple instructions as well as understand the content and purpose of the study.

Exclusion criteria:

1. Patients with severe dysphasia (either expressive or comprehensive) with inadequate communication.
2. Any additional medical or psychological condition affecting their ability to comply with the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Forearm's Assisted Range of Motion | Baseline
  Forearm's assisted range of motion is a measurement to identify how far the person's joints range can move in pronation-supination assisted by the motor-cable-driven system. The moving range will be recorded by the system and stored in computer
Wrist's Assisted Range of Motion | Baseline
  Wrist's Assisted range of motion is a measurement to identify how far the person's joints range can move in flexion/extension, and radial deviation/ulnar deviation with the assistance of motor-cable-driven system. The moving range will be recorded by the system and stored in computer.

SECONDARY OUTCOMES:
Upper limb Fugl-Meyer Assessment (FMA) | Baseline
  Introduction: Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale that are related to wrist and forearm component. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index.
  Scores: With the component of upper extremity (max 4 scores), wrist (max 10 scores), passive joint motion (max 8 scores) and joint pain (max 8 scores), the total or maximum scores is the sum of all the component which is 30 and the minimum is 0. The score for a normal person is 30 scores. The higher the score indicates the better the condition of the subject.
Motor Assessment Scale (MAS) | Baseline
  Introduction: Motor function that are related to wrist and forearm are measured using the Motor Assessment Scale. The Motor Assessment Scale (MAS) is a performance-based scale that was developed as a means of assessing everyday motor function in patients with stroke. In MAS, task 1 and 3 in the hand movement sub-component assessment were accessed (MAS-Hand), as the two task is the most related component to the tested movement.
  Score: The total or maximum scores is 2, and minimum scores is 0. In this scale, the higher the score indicates the better the condition of the subject. The score for a healthy person is 2.
Modified Ashworth Scale | Baseline
  Introduction: The spasticity level of wrist is measured by using Modified Ashworth Scale. It measures resistance during passive soft-tissue stretching. This measure will only measure the wrist component, as forearm component is not included in this scale.
  Scoring: The total or maximum scores for the subscale is 4 and the minimum is 0 score. Higher scores indicates the higher the tone, lower score indicates less tone. 0 score indicates normal tone and no increase in tone, while 4 scores indicate affected part rigid in flexion or extension. All the scores will be summed.
  Procedure: The measuring procedure starts by holding the elbow as straight as possible at forearm pronated. Then, the patient's wrist is moved from maximum possible flexion to maximum possible extension. The test is performed up tp maximum of 3 times to avoid the influence of the effect of stretch.
Forearm's Active Range of Movement | Baseline
  Forearm's active range of motion is a measurement to identify how far the person's joints range can move in pronation-supination by moving with their own effort. The moving range will be recorded by the system and stored in computer.
Forearm's Passive Range of Motion | Baseline
  Forearm's passive range of motion is a measurement to identify how far the person's joints range can move in pronation-supination directed by a person manually. The moving range will be recorded by the system and stored in computer.
Wrist's active range of motion | Baseline
  Wrist's active range of motion is a measurement to identify how far the person's joints range can move in flexion/extension, and radial deviation/ulnar deviation by moving with their own effort. The moving range will be recorded by the system and stored in computer.
Wrist's Passive Range of Motion | Baseline
  Wrist's passive range of motion is a measurement to identify how far the person's joints range can move in flexion/extension, and radial deviation/ulnar deviation directed by a person manually. The moving range will be recorded by the system and stored in computer.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong